CLINICAL TRIAL: NCT07107503
Title: 10 Years' Follow-up Results of Ultrasound-guided Radiofrequency Ablation Versus Surgery for Low-risk Papillary Thyroid Micro-carcinoma
Status: Completed | Type: Observational
Sponsor: Yi Mao (Other)
Responsible Party: Sponsor-Investigator, Yi Mao, clinician, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: ChinaPLAGH202506
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Papillary Thyroid Microcarcinoma; Radiofrequency Ablation; Surgical Resection; Long-term Outcomes
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radiofrequency ablation
  Interventions: Procedure: Radiofrequency ablation alone
- surgical resection
  Interventions: Procedure: surgical resection

INTERVENTIONS:
Procedure: Radiofrequency ablation alone — RFA was performed by four US physicians with ≥ 10 years of experience in in-terventional US. Before ablation, the patients were placed in the supine position with the neck extended, and local anesthesia was administered with lidocaine (1%). RFAs were performed using the hydro-dissection, trans-isthmic and moving-shot techniques according to previously published guidelines. Ablation was terminated when the target tumor changed to a transient hyperechoic zone. Contrast-enhanced US (CEUS) was performed immediately after ablation to evaluate the ablation area. The presence of complications during or after thermal ablation and corresponding treatments was carefully evaluated. All patients were closely observed for 1-2 h after ablation in the hospital.
  Groups: Radiofrequency ablation
Procedure: surgical resection — SR was performed under general anesthesia by surgeons with>15 years of expe-rience in thyroid surgery. The decision to perform total thyroidectomy or lobectomy was made by individual surgeons and patients, based on patient preferences in consu
  Groups: surgical resection

SUMMARY:
Papillary thyroid micro-carcinoma (PTMC) generally demonstrates favorable prognosis. However, the potential risk of disease progression requires careful therapeutic consideration. Radiofrequency ablation (RFA) has garnered attention as a minimally invasive treatment option for patients with PTMC who choose to decline both surgical resection (SR) and active surveillance. However, comprehensive comparative studies evaluating RFA versus surgery regarding long-term oncological efficacy, quality-of-life, and cost-effectiveness in multicenter cohorts remain warranted. To compare the oncological outcomes, quality of life, and cost-effectiveness between RFA and SR for low-risk PTMC over 10 years' follow-up.

ELIGIBILITY:
Inclusion Criteria:

(a) PTC confirmed at FNA or CNB, with a maximum diameter of 1 cm; (b) no clinical or imaging evidence of extra-thyroidal extension (41-42) and no evidence of metastasis at preoperative ultrasonography (US) or neck computed tomography (CT), indicating clinical preoperative T1aN0M0; (c) no history of neck irradiation; (d) no prior thyroid surgery; (e) follow-up of ≥ 120 months.

Exclusion Criteria:

(a) severe coagulation disorder or organ failure, (b) evidence of an aggressive sub-type of PTC on biopsy, and (c) incomplete data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective multi-center study included patients with PTMC treated at four university-affiliated hospitals in China from April 2011 to December 2014.
Sampling Method: Non-Probability Sample
Enrollment: 757 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Tumor progression | The RFA group follow-ups were conducted at 1, 3, 6, 12, and every 12 months thereafter. The SR group follow-ups were conducted at 1, 6, 12 and every 12 months thereafter. All the patients finished at least 10-year follow-ups.
  Tumor progression included (1) local recurrence confirmed by biopsy, (2) new PTMC tumors confirmed by biopsy, (3) LN metastasis confirmed by biopsy, and (4) distant metastases.

IPD SHARING:
Plan to Share IPD: No